

## PARTICIPANT INFORMATION LETTER

**Title of study:** Language translation of knowledge mobilization resources: A randomized trial

**Principal Investigators:** Dr. Lisa Hartling

Department of Pediatrics,

Faculty of Medicine and Dentistry

University of Alberta

Edmonton, Alberta, Canada Email: <a href="mailto:hartling@ualberta.ca">hartling@ualberta.ca</a> Telephone: (780) 492-6124

Dr. Sarah Elliott

Department of Pediatrics,

Faculty of Medicine and Dentistry

University of Alberta

Edmonton, Alberta, Canada Email: <u>se2@ualberta.ca</u> Telephone: (780) 492-6124

Research Coordinator(s): Samantha Cyrkot

Chelseay Robles

**Invitation to Participate:** You are invited to participate in this research study because your first language is one of the following languages: French, Spanish, Ukrainian, Tagalog, Arabic, Chinese, or Punjabi. You are 18 years of age or older and live in Canada. You have either a computer or tablet. You also have Internet, email, and can read English.

Purpose of the Study: This study is being done to learn how people from different language communities understand and perceive knowledge mobilization (KM) resources translated into their first language. KM resources provide evidence-based information to help people make decisions about their health. The resource used in this study focuses on preventing post COVID-19 condition (PCC), also known as long COVID. Individuals do not need to have experience with PCC (or long COVID) to participate. Health organizations translate materials to ensure that everyone has access to clear and accurate health information, but we don't always know how well these translations meet the needs of different communities. By asking participants to review translated resources and give their feedback, we hope to better understand if the translation is clear, easy to read, and trustworthy. The results will help guide how translations are done in healthcare to better support diverse communities.

NCT ID not yet assigned Ethics ID: Pro00153815 Version 1. July 14, 2025 **Participation:** If you wish to participate in this study, please complete the online survey using the link provided. The survey will take approximately 10 to 15 minutes to complete. Once finished, click the "Submit" button at the end of the survey to record your responses. This is an anonymous survey; we will not collect identifying information through the survey link.

**Risks:** Potential risks and discomfort may include mild fatigue or frustration if participants find the text confusing or difficult to interpret. To minimize this, all materials have been pilot-tested for clarity and presented in a user-friendly format. You may withdraw from the study at any time without penalty.

**Benefits:** While there are no direct benefits to being in this study, you will read and learn about some recommendations for prevention of PCC. In addition, there is a scientific benefit. This study will contribute to our understanding of how best to translate KM resources and help researchers (and others) make health information more accessible and inclusive for diverse language communities in Canada.

Voluntary Participation: You are under no obligation to take part in the study. If you choose to participate, you may skip any question you do not wish to answer. Should you choose to withdraw partway through the electronic survey, simply close the link or exit the browser and no responses will be recorded or used. Since this is an anonymous survey, and we do not collect any identifiable information within the survey itself, once you click "Submit," your responses cannot be withdrawn. You will then be directed to a separate, unlinked form to enter your email address for the gift card. This ensures your survey responses remain anonymous.

Compensation (or Incentives): To thank you for your participation, you will receive a \$5 CAD Everything Gift Card. You are free to decline the incentive and may still participate in the study if you choose to. You will be eligible for the gift card once you complete and submit the survey by clicking the "Submit" button. If you do not complete the questionnaire, you will not be eligible for the gift card. To protect your anonymity, you will be asked to enter your first name and email address on a separate form at the end of the survey. This form is not connected to your survey responses.

Confidentiality and Anonymity: The information that you provide will remain strictly confidential. You will not be asked to give your name, email address, IP address, or any other identifying information as part of the survey itself. Therefore, your responses will remain anonymous. Should you choose to provide your first name and email to receive a gift card, they will be stored separately from the data set. Sometimes, by law, we may have to release your information with your name so we cannot guarantee absolute privacy. However, we will make every legal effort to make sure that your information is kept private. During research studies, it is also important that the data we get is accurate. For this reason, your data, including your name, may be looked at by people from the Research Ethics Board.

**Data Storage:** Data will be collected and managed using REDCap (Research Electronic Data Capture). REDCap has an extensive privacy policy (https://help.redcap.ualberta.ca/policy-procedure/privacy) that has been reviewed by the study team and determined suitable for this

NCT ID not yet assigned Ethics ID: Pro00153815 Version 1. July 14, 2025 study, and has been previously approved for research use at the University of Alberta. Data will be downloaded regularly and stored long-term on a secure server in the PI's faculty (Faculty of Medicine & Dentistry) at the University of Alberta. Upon completion of the study, the data will be archived on the Faculty of Medicine & Dentistry server. The Faculty of Medicine & Dentistry has secure network drives accessible by network linked, password-protected computers and the data will not be accessible to anyone outside of the research team. Identifiable electronic data (e.g., Gift card records) will be deleted at time of study completion. De-identified (anonymous) electronic data (questionnaire data) will be kept for 5 years. Should you choose to provide it, your email address and first name will be collected only for the purpose of sending the electronic gift card. No hard copies of the data files will be stored.

**Information about the Study Results:** The results of this study will not be shared directly to the participants. However, participants may access the published manuscript through public or institutional databases once it becomes available.

**Contact Information:** If you have any questions about the research now or later, please contact <a href="mailto:arche@ualberta.ca">arche@ualberta.ca</a>.

If you have any questions regarding your rights as a research participant, you may contact the University of Alberta Research Ethics Office at <a href="ethics@ualberta.ca">ethics@ualberta.ca</a> or +1(780)492-2615 and quote Ethics ID Pro00153815. This office is independent of the researchers.

**Consent:** By reviewing this letter and proceeding to complete and submit the survey means your consent to participate.

Please download a copy of this Study Information Letter to keep for your records and reference.

Thank you very much for taking part in this study.

NCT ID not yet assigned Ethics ID: Pro00153815 Version 1. July 14, 2025